CLINICAL TRIAL: NCT06036654
Title: A Multicenter Clinical Trial of Infrared Bioeffect System for the Treatment of Onychomycosis
Brief Title: Infrared Bioeffect System for the Treatment of Onychomycosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gao Xinghua (Other)
Collaborators: Jining Medical University (Other); Binzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Gao Xinghua, Vice President, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH20230410
Record Dates: First submitted 2023-08-24; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Hyperthermia
Keywords: hyperthermia; onychomycosis
MeSH Terms: conditions — Hyperthermia; Onychomycosis

STUDY DESIGN:
Intervention Model Description: Local hyperthermia for the Treatment of Onychomycosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local Hyperthermia for the Treatment of Onychomycosis (Experimental): (1) In months 0-2, local hyperthermia treatment was given once a week for 20 minutes each time, for a total of 9 times; (2) In months 2-4, at the same target lesion, once every 2 weeks, for a total of 4 times; (3) In months 4-6, once every 4 weeks, for a total of 2 times. The frequency of this course of treatment was 15 times lasting for 6 months, and follow-up ended 12 months from the first treatment.
  Interventions: Device: infrared thermotherapy instrument

INTERVENTIONS:
Device: infrared thermotherapy instrument — Only a single target nail was chosen among multiple onychomycosis to receive local hyperthermia treatment.

SUMMARY:
Onychomycosis is a common nail plate infection caused by dermatophytes, non-dermatophytic molds, and yeasts. The disease is difficult to achieve self-healing and predisposed to secondary bacterial infections. There are currently multiple medications that can be used for the treatment of onychomycosis. The limitations are high recurrence rate and high cost, time-consuming and drug interactions. Several FDA approved laser devices have been available for the treatment of onychomycosis since 2010. As an emerging physical therapy modality, laser and light have advantages including extensive applicable range, simple operation, less trauma, and it will not lead to generation of new resistant strains. Therefore, it has been popularized and applied in clinics, especially among elderly, immunocompromised patients, or those with liver and kidney dysfunction. Laser systems in the near-infrared spectrum (780 nm∼ 3,000 nm wavelength), which are commonly used in onychomycosis, exert their effect by direct heating of target tissues, but it can cause unbearable physical pain to the patient. Compared with laser, controllable infrared bioeffect system has the advantages of high safety, less trauma, and less pain. Reported in the literature, it has been observed that regression of distant, untreated skin lesions in patients treated locally with controllable infrared bioeffect system, especially in inflammatory skin diseases such as viral warts and sporotrichosis. The aim of the research is to evaluate the safety and efficacy of controllable infrared bioeffect system in treatment of onychomycosis.

DETAILED DESCRIPTION:
Mild local hyperthermia with a certain temperature range has been successfully used in treatment of some diseases. It has been applied in the treatment of some neoplasm, fungal and HPV infections. Previous studies regarding viral warts and sporotrichosis found that in patients with multiple lesions, the clearance of the target lesion is commonly followed by clearance of other distant lesions, a phenomenon suggesting that local hyperthermia could aid in establishing a specific immune response to eliminate pathogenic microorganisms. Investigators speculate that mild local hyperthermia was a potential treatment for onychomycosis. A prospective single arm clinical trial was conducted to evaluate the effectiveness and safety of mild local hyperthermia in the treatment of onychomycosis. Participants with onychomycosis with at least 2 nails involved were included. The treatment effect of the treated and the untreated nail onychomycosis was measured after 6 months and 12 months of initial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients between 18 and 70 years old.
2. Patients with Onychomycosis confirmed by clinic and microscopic examination or culture of fungi.
3. All subjects voluntarily joined this study with informed consents.
4. The subjects have good compliance and can cooperate with investigators follow-up study.

Exclusion Criteria:

1. The patients during the period of pregnancy or breastfeeding.
2. The systemic and topical antifungal drugs were withdrawn 1 year and 3 months before enrollment, respectively.
3. Patients who suffered from progressive disease, autoimmune, tumor diseases or other diseases adjudged by the investigator to be inappropriate for inclusion into the study.
4. Other conditions adjudged by the investigator to be inappropriate for inclusion into the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-02-24 (Estimated); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
Cure rate of the target nail | 6 months, 9 months and 12 months after the first treatment
  Clinical and mycological cure rate of the target nail at 6 months, 9 months and12 months after the first treatment

SECONDARY OUTCOMES:
Cure rate of non-targeted nail | 6 months, 9 months, 12 months after the first treatment
  Clinical and mycological cure rate of non-target nail at 6 months, 9 months and12 months after the first treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No